CLINICAL TRIAL: NCT02742623
Title: COSIMO Cancer Associated Thrombosis - Patient Reported Outcomes With Rivaroxaban. A Non-interventional Study on Patients Changing to Xarelto® for Treatment of Venous Thromboembolism (VTE) and Prevention of Recurrent VTE in Patients With Active Cancer.
Brief Title: A Non-interventional Study on Xarelto for Treatment of Venous Thromboembolism (VTE) and Prevention of Recurrent VTE in Patients With Active Cancer
Acronym: COSIMO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18137; XA1502 (Other: Company internal)
Record Dates: First submitted 2016-03-01; First posted 2016-04-19 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Venous Thrombosis and Pulmonary Embolism
Keywords: Cancer; Deep Venous Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Neoplasms | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban: Female and male patients with active cancer and treated with rivaroxaban after a diagnosis of DVT/ and/or PE
  Interventions: Drug: Rivaroxaban (Xarelto, BAY 59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY 59-7939) — Treatment with rivaroxaban for DVT and/ or PE and/ or prevention of recurrent DVT and PE according to local label

SUMMARY:
This study aims to collect patient reported outcomes and assess treatment satisfaction in active cancer patients treated with rivaroxaban for VTE (venous thromboembolism).

ELIGIBILITY:
Inclusion Criteria:

* Adult female and male patients with active cancer other than fully treated basal-cell or squamous-cell carcinoma of the skin (active cancer defined as the diagnosis or treatment of cancer in the previous < 6 months or recurrent or metastatic cancer)
* Patients that have been treated with standard of care anticoagulation (Low Molecular Weight Heparin / Vitamin K Antagonist) for treatment of DVT and/ or PE (index VTE event) and/ or prevention of recurrent DVT and PE for at least 4 weeks prior to inclusion in the study
* Patients for whom the decision was made to start rivaroxaban for treatment of DVT and/ or PE and/ or prevention of recurrent DVT and PE
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2
* Patients who are willing to participate in this study (signed informed consent)
* Patients who are available for follow-up with a life expectancy >6 months

Exclusion Criteria:

* The contra-indications according to the local marketing authorization must be considered
* Patients who developed an index VTE event despite chronic anticoagulant therapy
* Patients receiving apixaban, edoxaban or dabigatran or any investigational drug as the initial therapy for the index VTE event
* Patients participating in an investigational program with interventions outside of routine clinical practice with exception of oncology investigational trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients with active cancer and a diagnosis of DVT/ and/or PE after the decision for treatment with rivaroxaban
Sampling Method: Non-Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction burden score (ACTS) | At 4 weeks
  Patient reported treatment satisfaction will be assessed with regard to the Anti-Clot Treatment Scale (ACTS) burden score for the use of rivaroxaban for treatment of acute deep vein thrombosis (DVT) and pulmonary embolism (PE), and prevention of recurrent DVT and PE in patients with active cancer changing to this therapy.

SECONDARY OUTCOMES:
Preferences regarding the attributes of the anticoagulation medication options LMWH, VKA, rivaroxaban using DCE survey | Between 4 weeks and 3 months
  Discrete Choice Experiment (DCE) based preference of patients for rivaroxaban versus other anticoagulants in a semi-structured telephone interview
  LMWH: Low Molecular Weight Heparin; VKA: Vitamin K Antagonist
Change of ACTS score over time | At 3 months and 6 months
  To assess patient reported outcomes by means of the Anti-Clot Treatment Scale (ACTS) questionnaire
Patient's quality of life using the FACIT-Fatigue questionnaire | Up to 6 months
  To assess patient reported outcomes on quality of life using the FACIT-Fatigue questionnaire (Functional Assessment of Chronic Illness Therapy)
Type of index VTE (venous thromboembolism) event | At baseline
Date of index VTE event | At baseline
Type (trade name) of initial anticoagulation treatment | At baseline
Duration of initial anticoagulation treatment | At baseline
Reason for drug switch to rivaroxaban | At baseline
  Menu items: patient choice, physician choice, side effects, other
Planned duration of anticoagulation with rivaroxaban | At baseline
Actual duration of anticoagulation with rivaroxaban | Up to 6 months
Dosage of rivaroxaban | Up to 6 months
Reason for any potential dose adjustments during course of treatment with rivaroxaban | Up to 6 months
  Menu items: side effects, intervention, other
Reasons for any switch from rivaroxaban treatment | Up to 6 months
  Menu items: patient choice, physician choice, side effects, other
Reasons for permanent cessation of rivaroxaban treatment | Up to 6 months
  Menu items: patient choice, physician choice, side effects, other
TNM Staging (Clinical characteristics of cancer disease) | At baseline
  Assessment according to TNM (Tumor, Lymph Node and Metastases) classification. TNM is developed and maintained by the Union for International Cancer Control (UICC)
Primary site of cancer (Clinical characteristics of cancer disease) | At baseline
  Following Medical Dictionary for Regulatory Activities (MedDRA) coding system
Type of bleeding events | Up to 6 months
Number of bleeding events | Up to 6 months
Type of thromboembolic events | Up to 6 months
Number of thromboembolic events | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Multiple Locations, Australia
- Multiple Locations, Belgium
- Multiple Locations, Canada
- Multiple Locations, Denmark
- Multiple Locations, France
- Multiple Locations, Germany
- Multiple Locations, Italy
- Multiple Locations, Netherlands
- Multiple Locations, Spain
- Multiple Locations, United Kingdom

REFERENCES:
- [Result] Maraveyas A, Beyer-Westendorf J, Lee AY, Mantovani LG, De Sanctis Y, Abdelgawwad K, Fatoba S, Bach M, Cohen AT. Cancer-Associated ThrOmboSIs - Patient-Reported OutcoMes With RivarOxaban (COSIMO) - Baseline characteristics and clinical outcomes. Res Pract Thromb Haemost. 2021 Nov 30;5(8):e12604. doi: 10.1002/rth2.12604. eCollection 2021 Dec. PMID 34877446
- [Derived] Cohen AT, Maraveyas A, Beyer-Westendorf J, Lee AYY, Mantovani LG, Bach M; COSIMO Investigators. COSIMO - patients with active cancer changing to rivaroxaban for the treatment and prevention of recurrent venous thromboembolism: a non-interventional study. Thromb J. 2018 Sep 4;16:21. doi: 10.1186/s12959-018-0176-2. eCollection 2018. PMID 30186045
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/18137